CLINICAL TRIAL: NCT02653924
Title: The Comparison of Microbial Adherence to Various Sutures in Patients Undergoing Oral Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HadassahMC
Record Dates: First submitted 2016-01-07; First posted 2016-01-13 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Oral Surgical Procedures
Keywords: Suture; bacteria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- silk suture (Active Comparator): silk suture
  Interventions: Other: silk suture
- vicryl suture (Active Comparator): vicryl suture
  Interventions: Other: vicryl suture
- nylon suture (Active Comparator): nylon suture
  Interventions: Other: nylon suture
- polypropylene suture (Active Comparator): polypropylene suture
  Interventions: Other: polypropylene suture

INTERVENTIONS:
Other: silk suture — each treatment will include 4 types of suture (as described above). all subjects will receive the same types of sutures. treatment plan is NOT influenced by the suture material used.
  Other Names: selection of sutures
  Arms: silk suture
Other: vicryl suture — each treatment will include 4 types of suture (as described above). all subjects will receive the same types of sutures. treatment plan is NOT influenced by the suture material used.
  Other Names: selection of sutures
  Arms: vicryl suture
Other: nylon suture — each treatment will include 4 types of suture (as described above). all subjects will receive the same types of sutures. treatment plan is NOT influenced by the suture material used.
  Other Names: selection of sutures
  Arms: nylon suture
Other: polypropylene suture — each treatment will include 4 types of suture (as described above). all subjects will receive the same types of sutures. treatment plan is NOT influenced by the suture material used.
  Other Names: selection of sutures
  Arms: polypropylene suture

SUMMARY:
The final stage of any surgical procedure is suturing. Sutures have a vital rule in wound healing- they are responsible for flaps approximation, hemostasis and restoring function and esthetics.

Choosing the right suture is crucial especially in oral sites because of its unique anatomical features: the presence of saliva and the patient's everyday function- swallowing, talking, eating etc.

Sutures require certain physical properties such as tensile strength, dimensional stability, lack of memory, knot security and elasticity. One highly important quality is the ability to prevent or reduce bacterial adhesion and by that to prevent secondary infection. There are many kinds of sutures in the market- none of which contains all the ideal features.

The aim of the study is to compare the amount of bacterial adhesion to different kinds of sutures in patients undergoing periodontal surgery.

DETAILED DESCRIPTION:
The participates in the study are scheduled to go oral surgery: dental implantation, Guided bone regeneration, resective periodontal surgery, sinus elevation (both crestal or lateral).

All participates will sign an informed consent form and under the institutional ethics committee approval will go to through the operation.

Each surgery will include at least 4 Simple Interrupted Suture with even spacing of 5 mm from each other in the scheduled for operation and without changing the original treatment plan. Incision location is in the area of surgery and not in a distinct location. The four sutures that will be used are: silk, vicryl, nylon and polypropylene.

At suture removal, after 10 days, all sutures will be collected in a sterile tube containing PBS solution. Within 3 hours, the samples will be sowed on two blood agar media plates. One plate will be aerobic condition and the other in an-aerobic condition. After one week, the number of colonies will use to calculate the CFU- colony-forming units.

ELIGIBILITY:
Inclusion Criteria:

* Patients designated for oral surgery with the possibility to perform at least 4 sutures, 5mm apart. The surgery will take place at the periodontology department, Dental faculty, Hadassah medical center.
* Patients willing to participate in the study and sign an informed concerned form
* Patients without systemic illness

Exclusion Criteria:

* Diabetes, heart disease, immune deficiency, thrombocytopenia\ coagulation enzymes deficiency
* Chronic alcohol consumption\ drug user
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
bacterial counts on blood agar plates from each suture will be quantified in CFU (colony-forming units) and expressed as total bacteria/suture | Outcome measure will be assessed 10 days after sample incubation for the different sutures obtained from each study participate
  CFU from all four different sutures (silk, vicryl, nylon and polypropylene sutures) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Dudu Polak, DMD, Principal Investigator — Department of Periodontology, Hadassah Medical Center, Jerusalem

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banche G, Roana J, Mandras N, Amasio M, Gallesio C, Allizond V, Angeretti A, Tullio V, Cuffini AM. Microbial adherence on various intraoral suture materials in patients undergoing dental surgery. J Oral Maxillofac Surg. 2007 Aug;65(8):1503-7. doi: 10.1016/j.joms.2006.10.066. PMID 17656275
- [Result] Selvig KA, Biagiotti GR, Leknes KN, Wikesjo UM. Oral tissue reactions to suture materials. Int J Periodontics Restorative Dent. 1998 Oct;18(5):474-87. PMID 10093524
- [Result] Grigg TR, Liewehr FR, Patton WR, Buxton TB, McPherson JC. Effect of the wicking behavior of multifilament sutures. J Endod. 2004 Sep;30(9):649-52. doi: 10.1097/01.don.0000121617.67923.05. PMID 15329570